CLINICAL TRIAL: NCT00854087
Title: A Phase II, Randomized, Placebo-Controlled, Double-Blind, Multi-Center Study to Assess the Antifibrotic Activity of Fuzheng Huayu in Chronic Hepatitis C Patients With Hepatic Fibrosis
Brief Title: Assess the Antifibrotic Activity of Fuzheng Huayu in Chronic Hepatitis C Patients With Hepatic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tarek Hassanein (Individual)
Collaborators: Shanghai Sundise Traditional Chinese Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Tarek Hassanein, Medical Director, SCTI Research Foundation
Organization: SCTI Research Foundation (Individual)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Fuzheng Huayu S-USIIT-01 Study
Record Dates: First submitted 2009-02-26; First posted 2009-03-02 (Estimated); Results first posted 2014-06-18 (Estimated); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Chronic Hepatitis C Infection
Keywords: Hepatitis C Virus; HCV; Herbal treatment; Herbs; San Diego; Non responder; Relapser; Treatment failure; Antifibrotic; Anti-fibrotic; Fibrosis; Failure of previous Interferon based therapy; Refuse Interferon based therapy; Intolerance to Interferon; Male or female 18-70 years of age
MeSH Terms: conditions — Hepatitis C; Fibrosis | interventions — fuzheng huayu; ping gan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fuzheng Huayu (Active Comparator): Pill with Fuzheng Huayu
  Interventions: Drug: Fuzheng Huayu
- Placebo (Placebo Comparator): Pill without Fuzheng Huayu (sugar pill)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fuzheng Huayu — The subjects will be taking 2 tablets three times a day for 48 weeks.
  Other Names: Gan Ping; 319 Recipe; FZHY
  Arms: Fuzheng Huayu
Drug: Placebo — The subjects will be taking 2 tablets three times a day for 48 weeks.
  Arms: Placebo

SUMMARY:
Current treatment of chronic liver disease relies upon removing the primary insult to the liver (e.g., alcohol) or treating the underlying viral infection (HBV, HCV, etc.). However, in the case of hepatitis C, a significant number of individuals will not clear the virus with current approved standard antiviral therapy, leaving them no options to manage their hepatic fibrosis, which can progress to cirrhosis and ultimately hepatocellular carcinoma (HCC).

Fuzheng Huayu has been used in numerous studies in China and has been found to have a satisfactory prophylaxis effect on the chronic liver injury and formed liver fibrosis in rats and humans. In addition, it enhances the degradation of liver fibrosis and protects hepatocytes from injury and death, manifesting as decreasing of ALT and AST, and enhancement of albumin level. In addition, preliminary studies indicate that the Fuzheng Huayu has a good safety and tolerability profile with promising efficacy.

The number of patients failing Interferon based therapy (i.e. not achieving SVR) is increasing. There are no approved standard of care treatment options for this population nor for patients who are intolerant or unwilling to receive Interferon; thus they are at higher risk for the progression of fibrosis. Moreover, there are no approved therapies to treat hepatic fibrosis, but basic research is exploring the pathophysiological mechanisms. Fuzheng Huayu is easy to administer, with a good safety and efficacy profile against fibrosis. Therefore, the investigators propose to further study the safety and efficacy profile of Fuzheng Huayu in a randomized, placebo-controlled, double blind study in Chronic Hepatitis C patients with hepatic fibrosis who have failed prior anti-HCV therapy or are intolerant or refuse Interferon based therapy.

The primary objective of this study is to establish the safety and efficacy of Fuzheng Huayu treatment in chronic hepatitis C subjects who have failed prior anti-HCV therapy or cannot receive or refused Interferon based therapy in improving liver fibrosis.

ELIGIBILITY:
Main Inclusion Criteria:

1. Male or female 18-70 years of age.
2. Chronic hepatitis C infection based on documented history of a positive serum anti-HCV antibody test and/or detectable levels of HCV RNA ≥ 50 IU/mL.
3. Failure to achieve sustained Virologic response (SVR) with previous Interferon based therapy or subjects who refuse Interferon based therapy or are intolerant to Interferon.
4. All subjects enrolling in the study and all fertile or potentially fertile sexual partners of subjects must be using two reliable forms of effective contraception during the study unless a study participant/partner is surgically sterile or postmenopausal.

Main Exclusion Criteria:

1. Subjects with any history of decompensated liver disease, including but not restricted to portal hypertension as manifested by gastroesophageal varices, variceal bleeding, ascites, or encephalopathy or a hepatic mass lesion suspicious for hepatocellular carcinoma (HCC).
2. Liver histology consistent with any other co-existing cause of chronic liver disease (apart from fatty liver).
3. Subjects who have been treated for HCV infection within 6 months before Screening.
4. Subjects who have been on any experimental protocol or therapy within 28 days before Screening.
5. Known HIV infection.
6. Chronic hepatitis B infection
7. Uncontrolled diabetes.
8. Unstable or uncontrolled thyroid disease
9. Uncontrolled seizures disorder.
10. History of malignant cancer within the last 5 years with the exception of localized basal or squamous cell carcinoma.
11. Alcohol and/or drug abuse within the past year.
12. Pregnant or lactating women or women who plan to become pregnant during the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2010-08; Primary Completion 2013-04 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Hassanein, MD, Principal Investigator — SCTI Research Foundation
Locations (8):
- United States (8):
  - SCTI Research Foundation, Coronado, California
  - VA Palo Alto HCS, Palo Alto, California
  - Huntington Medical Research Institutes, Pasadena, California
  - UC Davis Health System, Sacramento, California
  - Southern California Liver Centers, San Clemente, California
  - Advanced Medical Research Center, Port Orange, Florida
  - St. Luke's Advanced Liver Therapies, Houston, Texas
  - University of Utah HSC, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fuzheng Huayu | Placebo
Started | 59 | 59
Completed | 40 | 40
Not Completed | 19 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fuzheng Huayu | Placebo | Total
Number analyzed (Participants) | 59 | 59 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (6.72) | 55.1 (8.61) | 55.3 (7.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 23 | 48
  Male | 34 | 36 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 9 | 14
  Not Hispanic or Latino | 54 | 50 | 104
  Unknown or Not Reported | 0 | 0 | 0
HCV Genotypes [Number; unit: participants]
  1 | 48 | 52 | 100
  2 | 4 | 1 | 5
  3 | 6 | 5 | 11
  4 | 1 | 0 | 1
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety of Fuzheng Huayu Treatment in Chronic Hepatitis C Subjects Who Have Failed Prior Anti-HCV Therapy or Cannot Receive or Refused Interferon Based Therapy.
Description: Safety will be evaluated through the changes in vital signs, physical examinations, adverse events, concomitant medication assessments as well as laboratory tests.
Time Frame: Baseline to Week 60
Population: Number of participants randomized and who received at least one dose of Fuzheng Huayu or Placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Fuzheng Huayu | Placebo
Number analyzed (Participants) | 59 | 59
Participants
  Number of participants who experienced at least one adverse event | 55 | 55
  Number of participants who experienced at least one adverse event related to study drug | 42 | 38
  Number of participants who experienced at least one serious adverse event | 7 | 10
  Number of participants who experienced at least one serious adverse event related to study drug | 0 | 1
  Number of participants who had worsening of white blood cell count from baseline to week 48 | 42 | 45
  Number of participants who had worsening of Platelets count from baseline to week 48 | 42 | 45
  Number of participants who had worsening of liver enzymes from baseline to week 48 | 43 | 45

2. Primary Outcome: Efficacy of Fuzheng Huayu Treatment in Chronic Hepatitis C Subjects Who Have Failed Prior Anti-HCV Therapy or Cannot Receive or Refused Interferon Based Therapy.
Description: Efficacy of Fuzheng Huayu treatment was assessed through the change in liver fibrosis stage from the assessment before (pre) and after (post) study drug. The liver fibrosis staging system used was the Ishak scale. The Ishak liver fibrosis score ranges from 0 indicating no fibrosis to 6 indicating cirrhosis.
  "Fibrosis improved" was defined as a lower post study drug Ishak score, by at least 1 point, from pre-study drug assessment of the liver fibrosis e.g. if a pre study drug Ishak score of 4 and then a post study drug Ishak score of 3 or lower.
  "Fibrosis did not change" was defined as having the same Ishak score before and after study drug assessments e.g. if a pre study drug Ishak score of 4 and then a post study drug Ishak score of 4.
  "Fibrosis worsened" was defined as a higher post study drug Ishak score, by at least 1 point, from pre-study drug assessment of the liver fibrosis e.g. if a pre study drug Ishak score of 4 and then a post study drug Ishak score of 5 or higher.
Time Frame: Baseline to Week 48
Population: Participants who at least took one dose of study drug (Fuzheng Huayu or Placebo), were more than 80% compliant with study drug and had a pre and post study drug biopsy with an evaluable Ishak fibrosis score. Participants had ALT <300 and a BMI <40.
Measure: Number; unit: participants
Arm/Group | Fuzheng Huayu | Placebo
Number analyzed (Participants) | 38 | 43
participants
  Fibrosis improved | 9 | 13
  Fibrosis did not change | 18 | 12
  Fibrosis worsened | 11 | 18

ADVERSE EVENTS:
Time Frame: Study duration (screening through last study visit)
Arm/Group | Fuzheng Huayu | Placebo
Serious Adverse Events (participants affected / at risk) | 7/59 | 10/59
Other Adverse Events (participants affected / at risk) | 55/59 | 55/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fuzheng Huayu (N=59) | Placebo (N=59)
Sinus Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Bowel Obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Alcohol Rehabilitation (Social circumstances) | 0 (0) | 1 (1)
Atypical Chest Pain (General disorders) | 1 (1) | 0 (0)
T-12 Compression (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Opiod Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pleomorphic Rhabdomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Transverse Myelilitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ovarian Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute Hepatitis (Infections and infestations) | 0 (0) | 1 (1)
Hypokalemia/Hyponatremia/Nausea/Vomiting (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fuzheng Huayu (N=59) | Placebo (N=59)
Gastrointestinal disorders such as nausea (Gastrointestinal disorders) | 39 (84) | 30 (75)
General disorders such as fatigue (General disorders) | 27 (44) | 21 (27)
Infections such as urinary tract infection (Infections and infestations) | 24 (26) | 20 (34)
Respiratory such as cough (Respiratory, thoracic and mediastinal disorders) | 20 (36) | 24 (58)
Nervous system disorders such as headache (Nervous system disorders) | 20 (46) | 21 (35)
Psychiatric disorders such as depression (Psychiatric disorders) | 15 (20) | 15 (23)
Skin and subcutaneous system disorders such as rash (Skin and subcutaneous tissue disorders) | 14 (17) | 13 (19)
Injury, posioning and procedural complications such as muscle strain (Injury, poisoning and procedural complications) | 10 (11) | 12 (14)
Investigations such as liver biopsy (Investigations) | 6 (6) | 8 (8)
Surgical and medical procedures such as knee surgery (Surgical and medical procedures) | 6 (9) | 8 (8)
Metabolism and nutrition disorders such as decreased appetite (Metabolism and nutrition disorders) | 5 (8) | 5 (6)
Renal and urinary disorders such as nocturia (Renal and urinary disorders) | 7 (8) | 2 (2)
Vascular disorders such as hypertension (Vascular disorders) | 2 (2) | 5 (7)
Cardiac disorders such as tachycardia (Cardiac disorders) | 2 (2) | 4 (4)
Eye disorders such as dry eye (Eye disorders) | 3 (3) | 3 (3)
Immune system disorders such as rhinitis allergy (Immune system disorders) | 3 (3) | 3 (3)
Ear disorders such as vertigo (Ear and labyrinth disorders) | 3 (3) | 1 (1)
Neoplasms such as ovarian cysts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Reproductive system disorders such as erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 2 (3)
Endocrine disorders (hypothyroidism) (Endocrine disorders) | 0 (0) | 1 (1)
Hepatobiliary disorders (acute cholecistitis) (Hepatobiliary disorders) | 1 (1) | 0 (0)
Social circumstances (alcohol rehabilitation) (Social circumstances) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less